CLINICAL TRIAL: NCT03220828
Title: Evaluation of Technology-Based Stress Reduction Techniques Prior to Vascular Access
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Samuel Rodriguez, Assistant Professor,Department of Anesthesiology, Perioperative and Pain Medicine, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 40232
Record Dates: First submitted 2017-06-01; First posted 2017-07-18 (Actual); Last update posted 2019-04-16 (Actual); Status verified 2019-04

CONDITIONS: Stress, Emotional
MeSH Terms: conditions — Stress, Psychological

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): The control group will be provided standard of care, which is no use of technologies.
- Intervention Group VR (Experimental): Interventional arm will use technology based distractions (Virtual Reality)
  Interventions: Behavioral: Technology Based Distractions

INTERVENTIONS:
Behavioral: Technology Based Distractions — Technology based distractions (VR headsets)
  Arms: Intervention Group VR

SUMMARY:
Preprocedural, preoperative, and prevascular access anxiety in pediatric patients has been previously shown to increase the likelihood of family stressors, postoperative pain, agitation, sleep disturbances, and negative behavioral changes. The purpose of this study is to determine if a non-invasive distracting devices (Virtual Reality headset) is more effective than the standard of care (i.e., no technology based distraction) for preventing anxiety before vascular access among hospitalized children undergoing vascular access prior to anesthesia, procedures, surgery, blood draws, port access, or peripheral IV placement. The anticipated primary outcome will be reduction of child's anxiety during and after vascular access.

DETAILED DESCRIPTION:
Anxiety among children undergoing vascular access is common. Not only is high anxiety traumatic, but research indicates that high anxiety in children before surgery leads to adverse outcomes such as increased pain and analgesics requirements, delayed hospital discharge, and maladaptive behavioral changes. Treating anxiety may decrease any of these undesirable behaviors.

In this study, investigators hope to determine if technology based distractions (VR headsets) are more effective than standard care for preventing high anxiety before vascular access. As a secondary aim of the study, we seek to determine if the use of technology based distraction will result in higher parent and patient satisfaction, decreased fear, and increased compliance, while monitoring for side-effects of the intervention.

ELIGIBILITY:
Inclusion Criteria:

1. be between ages of 7-18 years of age
2. have comprehension of instructions in the English language
3. have parental consent
4. Pediatric patient must be undergoing non-emergent vascular access at Lucile Packard Children's Hospital in one of the 6 previously defined care areas (please see study design in Section 16).
5. Children who are normally healthy (ASA I) or have a mild systemic disease (ASA II,III)-

Exclusion Criteria:

1. Significant cognitive impairment/developmental delays per parental report or H&P.
2. Children with ASA IV (severe systemic disease that is a constant threat to life) or ASA V (unstable patients not expected to survive >24hours or without the operation)
3. H/o severe motion sickness, nausea, seizures

Ages: 7 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 220 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2019-03-31 (Actual); Study Completion 2019-03-31 (Actual)

PRIMARY OUTCOMES:
Change in Pain Score | immediately post vascular access minus baseline
  Peak Pain Score minus Baseline Pain Score(0-10)

SECONDARY OUTCOMES:
Fear Score | immediately post vascular access minus baseline
  Fear Faces
Family Satisfaction | Immediatly Post Vascular Access
  Family Satisfaction Survey
Patient Satisfaction | Immediately Post Vascular Access
  Patient Satisfaction Survey
Patient Compliance | At the time of Vascular Access
  Modified Induction Compliance Checklist
Adverse Events | At the time of Vascular Access
  Negative outcomes such as nausea, headache

CONTACTS AND LOCATIONS:
Overall Officials: Samuel Rodriguez, MD, Principal Investigator — Stanford University
Locations (1):
- Lucile Packard Children's Hospital at Stanford, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: Undecided